Effect of Longitudinal Care in Primary Health Care: An Analysis from the Patient's Perspective

February 2024

Acronym: CUALIPRIM

## **Informed Consent Form**

| <b>Project Title:</b> Longitudinality in Primary Health Care: an analysis from the patient's perspective. | |
|---|---|
| Surname and Name: | |
| ID Number (DNI / NIE): | |
| Health Card Number (NUHSA): | |
| PROFESSIONALS INVOLVED IN THE INFO | RMATION AND/OR CONSENT PROCESS |
| The following professionals declare that they have in the project: | ve provided the information related to participation |
| Surname and Name – Date – Signature | |
| CONSENT | |
| I, Mr./Ms I have read and understood the Information Shee | , declare under my responsibility that et, of which I have been given a copy. |
| I have received sufficient information regarding my personal data | my participation in the project, regarding the use of |
| and associated information. I have been able to a speak with the designated professional, who has | ask questions about the information received and |
| I understand that my participation is voluntary. | |
| I understand that all my data will be treated confined of 5 December on Personal Data Protection and I understand that I may withdraw from the study | $\varepsilon$ $\varepsilon$ |
| - Whenever I wish. | |
| <ul><li>Without having to provide any explanation.</li><li>Without this affecting my medical care.</li></ul> | |
| | ressed in an anonymised manner (the samples/data and my identity has been irreversibly removed). |
| I am aware that I may revoke, at any time, the co<br>(When data or samples are anonymised, this poin | |
| In, on the | day of20 |
| THE DONOR | PARTICIPANT LEGAL REPRESENTATIVE (only in cases of incapacity) |
| Signature: | Signature: |

## **EXAMPLE OF REVOCATION OF INFORMED CONSENT** I, Mr/Ms. with ID number ..... declare that: I have read the Information Sheet and the Revocation of Informed Consent document 1. provided to me. 2. I have discussed and clarified any doubts regarding my revocation with Dr. 3. I hereby revoke the consent previously granted, which becomes invalid from this moment onwards. My revocation is: □ Total □ Partial. Please specify: Signature:

## Regarding family members / guardians / legal representatives:

| The patient Mr./Ms | | , with ID | |
|---|---|---|---|
| number | , does not have decision | on-making capacity at this time. | |
| Therefore, Mr./Ms | ••••• | , with ID | |
| numberpreviously granted, which b | , 0 | moment onwards. | nsent |
| In, | on the day of | 20 | |
| Signature: | | | |

## APPLICABLE REGULATIONS

- Law 14/2007, of 3 July, on Biomedical Research.
- Law 41/2002, of 14 November, basic law regulating patient autonomy and rights and obligations regarding clinical information and documentation.
- Royal Decree 1716/2011, of 18 November, establishing the basic requirements for the authorisation and operation of biobanks for biomedical research purposes and for the processing of human biological samples, and regulating the National Registry of Biobanks.
- Regulation (EU) 2016/679 of the European Parliament and of the Council, of 27 April 2016, on the protection
  of natural persons with regard to the processing of personal data and the free movement of such data (General
  Data Protection Regulation).
- Organic Law 3/2018, of 5 December, on Personal Data Protection and guarantee of digital rights.